CLINICAL TRIAL: NCT06095609
Title: The Implementation of Early Mobilization and Chest Physiotherapy on Weaning Rate of Prolong Weaning Patients. A Retrospective Study
Brief Title: The Implementation of Early Mobilization and Chest Physiotherapy on Weaning Rate of Prolong Weaning Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYGH111002
Record Dates: First submitted 2022-06-20; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-09

CONDITIONS: Prolonged Weaning, Early Mobilization, Chest Physiotherapy
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: The study retrospectively reviewed the medical record from the medical team. Patients before 2019/01/01 who didn't receive physiotherapy are regarded as control group. Patients after 2019/01/01 are assigned to the experiment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization plus chest physiotherapy (Experimental): Physiotherapy program comprised two parts early mobilization and CPT. They could be divided into different levels depended on patients' ability. In terms of the levels of early mobilization, first level was defined as patients who could only receive passive patterns of exercise. Second level would be executed to patient who could only take exercise on the bed or with back support. Third level would be implemented when patients could advance to receive physiotherapy beside the bed without support. The eventual level would be conducted when patients was able to leave beds by their own. In line with chest physiotherapy, level I was defined as patients who could only receive passive lung hygiene protocol. Level II would be executed when patient can control their breath and cough by their own. Level III would be implemented when patient can maintain their body steadily and finish the chest physiotherapy protocol.
  Interventions: Other: Early mobilization plus chest physiotherapy
- Routine care (No Intervention): no physiotherapy involved

INTERVENTIONS:
Other: Early mobilization plus chest physiotherapy — Early mobilization:early mobilization has been confirmed its positive effectiveness on cutting down the MV use days and mortality rate, attenuating the side effect such as muscle strength loss and functional activity dysfunction resulting from ICU acquired weakness among the patients with mechanical ventilation.
  Chest physiotherapy:a common technique to reduce the respiratory complications in ICU, has been proved certain positive influence on airway clearance and hospital lengths of stay.
  Arms: Early mobilization plus chest physiotherapy

SUMMARY:
Weaning from mechanical ventilator is essential to liberate patients to normal life. Prolong weaning is defined as failure of 3 times spontaneous breath trial (SBT) and requiring more than 7 days weaning from mechanical ventilation after first SBT. higher unsuccessful rate of extubation and higher mortality rate. Possible reasons to cause prolong weaning could be attributed to intensive care unit acquired weakness (ICU-AW) and poor lung hygiene. In order to solve these two problems and increase the weaning rate, early mobilization (EM) and chest physiotherapy (CPT) are considered as possible strategy to attain the goal. According to previous articles, lacking of control group and small sample size made it difficult to confirm the true effect of EM and CPT on prolong weaning patients. Thus, the aims of this articles are discussing the influence from EM with CPT on weaning rate and other hospitalization outcomes with larger sample sizes and control group.

ELIGIBILITY:
Inclusion Criteria:

* The subjects' data which met the inclusion criteria are: 1. Age>20 2. Patient with or without 3. Patient who met the criteria of received physiotherapy (Figure 1.) 4. No usage of life support device such as ECMO and so on. 5. Continuous mechanical ventilator use over 21 days.

Exclusion Criteria:

* The exclusion criteria are 1. Patients diagnosed as brain death 2. Patients who were ventilator dependent before admission 3. Patients who were against advice discharge under critical condition. 4. Patients received emergency intervention during course. 5. Patient who didn't meet the criteria of received physiotherapy (Figure 1.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
Weaning success rate | up to 6 weeks in respiratory care center
  Weaning success was defined as patients being free from MV or BiPAP for 5 days based on Taiwan

SECONDARY OUTCOMES:
RCC mortality rate | up to 6 weeks in respiratory care center
  the mortality rate of respiratory care center
hospital mortality rate | up to 6 weeks in respiratory care center
  the mortality rate during the hospital course
discharge to home rate | after 6 weeks in respiratory care center
  The rate of going home after discharge
total mechanical ventilator use | up to 6 weeks in respiratory care center
  The days of mechanical use during the admission time
RCC days of stay | up to 6 weeks in respiratory care center
  The days staying in respiratory care center
total hospital days of stay | up to 10 weeks in the hospital
  The days staying in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyaun General Hospital, Ministry of Wealth and Health, Taoyuan District, Taoyuan Dist., Taiwan